CLINICAL TRIAL: NCT05374343
Title: A Phase I Study of the Pharmacokinetics/Pharmacodynamics and Safety of Rongliflozin in Chinese Subjects With Type 2 Diabetes With Normal Renal Function and Mild to Moderate Renal Impairment
Brief Title: A Study of the Pharmacokinetics, Pharmacodynamics, and Safety of Rongliflozin in Type 2 Diabetic Subjects With Renal Impairment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DJT1116PG-DM-106
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A and C (normal kidney function) (Active Comparator): Each subject will receive a single dose of rongliflozin on Day 1
  Interventions: Drug: pyroglutamate rongliflozin capsules
- Group B (mild renal impairment) (Experimental): Each subject will receive a single dose of rongliflozin on Day 1
  Interventions: Drug: pyroglutamate rongliflozin capsules
- Group D (moderate renal impairment) (Experimental): Each subject will receive a single dose of rongliflozin on Day 1
  Interventions: Drug: pyroglutamate rongliflozin capsules

INTERVENTIONS:
Drug: pyroglutamate rongliflozin capsules — Subjects will receive one 50mg capsule orally (by mouth) on Day 1

SUMMARY:
To evaluate the pharmacokinetic characteristics of pyroglutamate rongliflozin capsules in type 2 diabetic subjects with normal renal function and mild to moderate renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients.
* The subject is willing to take effective contraceptive measures without a pregnancy plan within 4 weeks after signing the informed consent form to taking the test drug.
* When screening, 19.0 kg/m2 < or = body mass index (BMI) < or = 35.0 kg/m2.
* No hypoglycemic drugs have been used in the 4 weeks before the baseline period, or stable doses of hypoglycemic drugs are being used.
* No medications for other comorbidities or stable medication regimens within 4 weeks before the baseline period.
* In the screening period, 6.5% < or = glycosylated hemoglobin < or =11.0%, and fasting blood glucose < or = 13.9 mmol/L.
* Glomerular filtration rate (eGFR) > or = 90 mL/min/1.73m2 estimated according to the modified dietary trial for kidney disease (MDRD) formula (only applicable to patients with type 2 diabetes with normal renal function).
* Accompanied by mild or moderate renal impairment, the eGFR calculated according to the MDRD formula meets the following criteria: mild renal impairment: 60~89 mL/min/1.73m2, moderate renal impairment: 30~59 mL/min/ 1.73m2 (only for patients with type 2 diabetes with impaired renal function).
* Accompanied by mild or moderate renal impairment, accompanied by stable disease in the first 3 months of the baseline period (only applicable to patients with type 2 diabetes with renal impairment).

Exclusion Criteria:

* Known allergy to sodium-glucose cotransporter 2 (SGLT2) inhibitor drugs or related excipients.
* In the 3 months before screening, those who smoked more than 5 cigarettes per day on average or who could not give up smoking from signing informed consent to leaving the group.
* Have a history of alcoholism.
* Ingested any food or drink containing caffeine, xanthine, alcohol, grapefruit within 48 hours before taking the test drug.
* Those who donate blood or lose a lot of blood (>400 mL) within 3 months before taking the test drug, or have a history of blood transfusion within 1 month before screening, or plan to donate blood within 1 month after the end of the trial.
* Those who have taken the trial drug or such drugs within 1 month before taking the trial drug, or participated in the clinical trial of any drug or medical device within 3 months before screening.
* Those who have a positive urine drug screen or have a history of drug abuse or drug use in the past 5 years.
* The subject is breastfeeding or the serum pregnancy test result is positive.
* Subjects had undergone surgery within 1 month before screening, or major surgery was planned during the study period.
* Have severe mental illness or language barrier, unwilling or unable to fully understand and cooperate.
* History or evidence of other diseases, such as history of repeated urinary tract infections, poorly controlled high blood pressure, type I diabetes, urinary incontinence, etc.
* Abnormal laboratory tests, such as a) Alanine transaminase (ALT)/Aspartate aminotransferase (AST)>2.0×UNL and/or total bilirubin>1.5×UNL; b) hemoglobin <100 g/L; c) hepatitis B surface antigen positive, hepatitis C antibody positive, HIV antibody positive , Syphilis antibody positive.
* The researcher believes that the subject has any situation that may interfere with the interpretation of the pharmacokinetics, efficacy and safety data of this study.
* Subjects considered by the researcher to be unsuitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-02-13 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of rongliflozin | 0 hour（pre-dose） to 96 hours after administration
  Plasma concentrations of rongliflizin following the administration of a single dose of rongliflozin, the pharmacokinetic parameters for rongliflozin will be measured in varying degrees of kidney function.

SECONDARY OUTCOMES:
Change from baseline in 24-hour urine glucose excretion in varying degrees of kidney function | Day -1 (Baseline) to Day 5
  Change from baseline in 24-hour urine glucose excretion following the administration of a single dose of rongliflozin will be used to evaluate the pharmacodynamics of rongliflozin (ie, how the drug affects the body) in varying degrees of kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Feng, Doctor, Principal Investigator — West China Hospital; Zhenmei An, Master, Principal Investigator — West China Hospital
Locations (1):
- Ping Feng, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No